CLINICAL TRIAL: NCT01665105
Title: Study on the Effect of Electroacupuncture at Both Zusanli and at Both Yanglingquan Acupoints on Autonomic Nerve Modulating Cardiovascular Activity , and Skin Blood Flow and Skin Temperature
Brief Title: Study on the Effect of Electroacupuncture at Both Zusanli and at Both Yanglingquan Acupoints on Cardiovascular Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: DMR101-IRB2-101
Record Dates: First submitted 2012-07-20; First posted 2012-08-15 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Reaction of Autonomic Nervous System; Reaction of Acupuncture; Reaction of Blood Circulation
Keywords: Pulse Rate Variability; Skin Blood Flow; Skin Temperature; Electroacupuncture; Zusanli; Yanglingquan
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Zusanli Group (Experimental): electroacupuncture at both Zusanli on the leg, and record simultaneously the pulse rate variability as well as take the skin blood flow and skin temperature recordings at Hoku's and Zhongzhu's region of right hand.
  Interventions: Device: acupuncture
- Yanlingquan Group (Active Comparator): electroacupuncture at both Yanglingquan on the leg, and record simultaneously the pulse rate variability as well as take the skin blood flow and skin temperature recordings at Hoku's and Zhongzhu's region of right hand.
  Interventions: Device: acupuncture
- Sham Group (Sham Comparator): acupuncture without electrical stimulation at non-acupoint on the leg, and record simultaneously pulse rate variability as well as take the skin blood flow and skin temperature recordings at Hoku's and Zhongzhu's region of right hand.
  Interventions: Device: acupuncture

INTERVENTIONS:
Device: acupuncture — electroacupuncture at at Zusanli, electroacupuncture at Yanglingquan, and acupuncture at non-acupoint.

SUMMARY:
The purpose of this present study was to investigate the effect of electroacupuncture at both Zusanli and at both Yanglingquan acupoints on autonomic nerve modulating cardiovascular activity, and skin blood flow and skin temperature. The investigators use pulse rate variability to investigate autonomic nerve modulates cardiovascular function, and using distant skin blood flow and skin temperature recordings to investigate the relationship between the same names meridian of hand and foot.

DETAILED DESCRIPTION:
A total of 24 adult healthy volunteer were studied, they received the three sessions of sham electroacupuncture, electroacupuncture at Zusanli and electroacupuncture at Yanglingquan, respectively. Each session was divided into three periods of before electroacupuncture, electroacupuncture, and post electroacupuncture. Each period was 20 min in duration. The ahead 15 min of the period was the skin blood flow and skin temperature recordings at Hoku's and Zhongzhu's region of right hand; the final 5 min of the period was pulse rate variability recordings of left hand. The data was storage and analysis in a personal computer.

ELIGIBILITY:
Inclusion Criteria:

1. healthy volunteers without without cardiac disease, taking medications, smoking
2. before experiment, abstaining from caffeine, alcohol for 8 hours.
3. age between 20-40.

Exclusion Criteria:

1. volunteers with cardiac disease, taking medications, smoking
2. age greater than 40 or less than 20.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
From pulse wave, pulse rate variability and skin blood flow to measure cardiovascular activities with electroacupuncture at Zusanli and at Yanglingquan. | each period was 20 min in duration. The parameters of pulse wave, 5-min pulse rate variability were recorded at the end of each period.
  Each session was divided into three periods of before electroacupuncture, electroacupuncture, and post electroacupuncture. Each period was 20 min in duration. During each period, the final 5 min of the period was pulse rate variability recordings of left hand by ANSWatch(TS-0411 model). This data were storage as primary outcomes and analyzed in a personal computer.

SECONDARY OUTCOMES:
From skin blood flow and skin temperature to measure cardiovascular activities with electroacupuncture at Zusanli and at Yanglingquan. | each period was 20 min in duration. The parameters of skin blood flow and skin temperature were recorded at the end of each period.
  Each session was divided into three periods of before electroacupuncture, electroacupuncture, and post electroacupuncture. Each period was 20 min in duration. During each period, the ahead 15 min of the period was the skin blood flow and skin temperature recordings at Hoku's and Zhongzhu's region of right hand by Laser doppler blood flow monitor (Moor instruments DRT4 model). This data were storage as seconrdary outcomes and analyzed in a personal computer.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Liang Hsieh, professor, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan